CLINICAL TRIAL: NCT00598533
Title: Prospective, Randomized Trial of Rapamycin- and Zotarolimus-eluting Stents for the Reduction of Coronary Restenosis
Brief Title: Efficacy Study of Rapamycin- vs. Zotarolimus-Eluting Stents to Reduce Coronary Restenosis
Acronym: ISAR-TEST-5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE No. S02907
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual-DES (Experimental): Rapamycin + Probucol-eluting stent
  Interventions: Device: Rapamycin + Probucol-eluting stent (ISAR stent)
- ZES (Active Comparator): Polymer based Zotarolimus-eluting stent
  Interventions: Device: polymer based Zotarolimus-eluting stent (Endeavor Resolute)

INTERVENTIONS:
Device: Rapamycin + Probucol-eluting stent (ISAR stent) — due to randomization, Rapamycin- + Probucol-eluting stent will be implanted
  Other Names: ISAR stent
  Arms: Dual-DES
Device: polymer based Zotarolimus-eluting stent (Endeavor Resolute) — due to randomization, Zotarolimus-eluting stent with polymer will be implanted
  Other Names: Endeavor Resolute
  Arms: ZES

SUMMARY:
The purpose of this trial is to evaluate the efficacy of Rapamycin- and Zotarolimus-Eluting stents for the reduction of Coronary Restenosis

DETAILED DESCRIPTION:
This prospective, randomized trial will compare the efficacy and safety of a Rapamycin plus Probucol-eluting stent with a polymer based Zotarolimus-eluting stent. Patients with symptomatic coronary artery disease without cardiogenic shock who will undergo coronary angiography and willing to participate in the trial will receive a loading dose of 600mg clopidogrel at least 2 hours before the procedure. They will be randomized to receive one of the above mentioned stents.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% de novo stenosis located in native coronary vessels
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study
* In women with childbearing potential a negative pregnancy test is mandatory.

Exclusion Criteria:

* Target lesion located in the left main trunk.
* Target lesion located in the bypass graft.
* In-stent restenosis.
* Cardiogenic shock.
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Known allergy to the study medications: Clopidogrel, Rapamycin, Probucol, Zotarolimus, stainless steel or cobalt chrome.
* Inability to take clopidogrel for at least 6 months.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3002 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
A composite endpoint of cardiac death, myocardial infarction related to the target vessel or target lesion revascularisation | at one year

SECONDARY OUTCOMES:
Late luminal loss | at 6-8 months follow-up angiography
stent thrombosis | at one year

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - Medizinische Klinik, Klinikum rechts der Isar, München

REFERENCES:
- [Derived] Coughlan JJ, Aytekin A, Xhepa E, Cassese S, Joner M, Koch T, Wiebe J, Lenz T, Rheude T, Pellegrini C, Gewalt S, Ibrahim T, Laugwitz KL, Schunkert H, Kastrati A, Kufner S. Target and non-target vessel related events at 10 years post percutaneous coronary intervention. Clin Res Cardiol. 2022 Jul;111(7):787-794. doi: 10.1007/s00392-022-01986-4. Epub 2022 Feb 11. PMID 35147767
- [Derived] Koch T, Lenz T, Joner M, Xhepa E, Koppara T, Wiebe J, Coughlan JJ, Aytekin A, Ibrahim T, Kessler T, Cassese S, Laugwitz KL, Schunkert H, Kastrati A, Kufner S; Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting Versus Zotarolimus- Eluting Stents (ISAR-TEST 5) Investigators. Ten-year clinical outcomes of polymer-free versus durable polymer new-generation drug-eluting stent in patients with coronary artery disease with and without diabetes mellitus : Results of the Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol- and Zotarolimus-Eluting Stents (ISAR-TEST 5) trial. Clin Res Cardiol. 2021 Oct;110(10):1586-1598. doi: 10.1007/s00392-021-01854-7. Epub 2021 Jun 22. PMID 34156521
- [Derived] Kufner S, Ernst M, Cassese S, Joner M, Mayer K, Colleran R, Koppara T, Xhepa E, Koch T, Wiebe J, Ibrahim T, Fusaro M, Laugwitz KL, Schunkert H, Kastrati A, Byrne RA; ISAR-TEST-5 Investigators. 10-Year Outcomes From a Randomized Trial of Polymer-Free Versus Durable Polymer Drug-Eluting Coronary Stents. J Am Coll Cardiol. 2020 Jul 14;76(2):146-158. doi: 10.1016/j.jacc.2020.05.026. PMID 32646563
- [Derived] Harada Y, Colleran R, Kufner S, Giacoppo D, Rheude T, Michel J, Cassese S, Ibrahim T, Laugwitz KL, Kastrati A, Byrne RA; Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol- and Zotarolimus- Eluting Stents (ISAR-TEST 5) Investigators. Five-year clinical outcomes in patients with diabetes mellitus treated with polymer-free sirolimus- and probucol-eluting stents versus second-generation zotarolimus-eluting stents: a subgroup analysis of a randomized controlled trial. Cardiovasc Diabetol. 2016 Sep 1;15(1):124. doi: 10.1186/s12933-016-0429-y. PMID 27586678
- [Derived] Colleran R, Kufner S, Harada Y, Giacoppo D, Cassese S, Repp J, Wiebe J, Lohaus R, Lahmann A, Schneider S, Ibrahim T, Laugwitz KL, Kastrati A, Byrne RA; Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting Versus Zotarolimus-Eluting Stents (ISAR-TEST 5) Investigators. Five-year follow-up of polymer-free sirolimus- and probucol-eluting stents versus new generation zotarolimus-eluting stents in patients presenting with st-elevation myocardial infarction. Catheter Cardiovasc Interv. 2017 Feb 15;89(3):367-374. doi: 10.1002/ccd.26597. Epub 2016 Jul 5. PMID 27377301
- [Derived] Kufner S, Sorges J, Mehilli J, Cassese S, Repp J, Wiebe J, Lohaus R, Lahmann A, Rheude T, Ibrahim T, Massberg S, Laugwitz KL, Kastrati A, Byrne RA; ISAR-TEST-5 Investigators. Randomized Trial of Polymer-Free Sirolimus- and Probucol-Eluting Stents Versus Durable Polymer Zotarolimus-Eluting Stents: 5-Year Results of the ISAR-TEST-5 Trial. JACC Cardiovasc Interv. 2016 Apr 25;9(8):784-792. doi: 10.1016/j.jcin.2016.01.009. Epub 2016 Mar 23. PMID 27017366
- [Derived] Massberg S, Byrne RA, Kastrati A, Schulz S, Pache J, Hausleiter J, Ibrahim T, Fusaro M, Ott I, Schomig A, Laugwitz KL, Mehilli J; Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting Versus Zotarolimus- Eluting Stents (ISAR-TEST 5) Investigators. Polymer-free sirolimus- and probucol-eluting versus new generation zotarolimus-eluting stents in coronary artery disease: the Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting versus Zotarolimus-eluting Stents (ISAR-TEST 5) trial. Circulation. 2011 Aug 2;124(5):624-32. doi: 10.1161/CIRCULATIONAHA.111.026732. Epub 2011 Jul 18. PMID 21768546